CLINICAL TRIAL: NCT05888090
Title: The Effect of Position Given to Preterms After Feeding on Gastric Residual Volume, Abdominal Oxygenation and Fractional Oxygen Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, HANDE OZGORU, The Effect of Position Given to Preterms After Feeding on Gastric Residual Volume, Abdominal Oxygenation and Fractional Oxygen Extraction, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 14311537094
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Gastric Residual Volume; Abdominal Oxygenation; Fractional Oxygen Extraction; Positioning (Prone, Right Lateral and Semi-Elevated Supine Position)
Keywords: Preterm Infants; Positioning; Gastric Residual Volume; Abdominal Oxygenation; Fractional Oxygen Extraction
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Breastfed preterm neonates to be included in the study will be placed in 3 positions in a randomized crossover design. The order of the 3 positions that will be given to the babies in the research group will be determined by drawing lots and 3 intervention groups will be formed. Preterm newborns in each intervention group will be followed for two hours after feeding in all three positions: semi-elevated supine position, prone position, and right lateral position. Positions will be given to babies, taking into account the order of positions in each group. All positions will be applied once to each baby. Groups and position rankings according to the result of the draw:
  1. st group: Prone, right lateral and semi-raised supine position
  2. nd group: Semi-raised supine, prone and right lateral position
  3. rd group: Right lateral, semi-raised supine and prone position
  48 preterm newborns in the study group will be randomly assigned to these 3 intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Intervention Group 1 (Experimental)
  Interventions: Other: Prone, right lateral, and semi-elevated supine positions
- Intervention Group 2 (Experimental)
  Interventions: Other: Semi-elevated supine, prone, and right lateral positions
- Intervention Group 3 (Experimental)
  Interventions: Other: Right lateral, semi-elevated supine, and prone positions

INTERVENTIONS:
Other: Prone, right lateral, and semi-elevated supine positions — Each participant will be followed during three feedings and the prone, right lateral, and semi-elevated supine positions will be applied once.
  Arms: Intervention Group 1
Other: Semi-elevated supine, prone, and right lateral positions — Each participant will be followed during three feedings and the semi-elevated supine, prone, and right lateral positions will be applied once.
  Arms: Intervention Group 2
Other: Right lateral, semi-elevated supine, and prone positions — Each participant will be followed during three feedings and the right lateral, semi-elevated supine, and prone positions will be applied once.
  Arms: Intervention Group 3

SUMMARY:
This study is a PhD dissertation. In this study, the investigators aim to investigate the effects of three different positions after feeding on gastric residual volume, abdominal oxygenation using near infrared spectroscopy (NIRS), and fractional oxygen extraction values in preterm newborns.

DETAILED DESCRIPTION:
The Design of Research

This study was planned in a randomized crossover study design to evaluate the effects of three different positions on gastric residual volume, fractional oxygen extraction and abdominal oxygenation in clinically stable breastfed preterm newborns. The order of the 3 positions that will be given to the participants the research group will be determined by drawing lots and 3 intervention groups will be formed. The participants in each intervention group will be followed for two hours after feeding in all three positions: semi-elevated supine position, prone position, and right lateral position. Positions will be given to the participants, taking into account the order of positions in each group. All positions will be applied once to each participant. Groups and position rankings according to the result of the draw:

1. st group: Prone, right lateral, and semi-elevated supine position;
2. nd group: Semi-elevated supine, prone, and right lateral position;
3. rd group: Right lateral, semi-elevated supine, and prone position;

48 participants in the study group will be randomly assigned to these 3 intervention groups. In order to determine which participant will be in which group, the numbers from 1 to 48 were distributed to 3 groups through a program in the computer environment without repeating the number (https://www.randomizer.org/). Randomization is provided as follows.

Intervention group 1: 2.8,12,17,18,22,24,25,26,31,33,36,37,40,42,45; Intervention group 2: 1,3,5,10,14,16,19,20,27,28,29,30,32,34,43,44; Intervention group 3: 4,6,7,9,11,13,15,21,23,35,38,39,41,46,47,48;

Location and Time of Research Data of the research Istanbul Kartal Dr. Lütfi Kırdar City Hospital will meet at the Newborn Intensive Care Unit between July 2023 and July 2024. 2., 3., and the university hospital, which provides 4A level intensive care, consists of a total of 41 beds. It consists of 14 level beds, 3rd level 14 beds and 13 beds with 4A level.

Survey's Universe and Sampling After the necessary legal permits have been obtained in the universe of the research, (Ethical Board approval and institution permit ), Kartal Dr. at the time of the investigation. The preterm followed by the Lütfi Kırdar City Hospital Newborn Intensive Care Unit will create newborns.

The sample of the research is Eagle Dr. Lütfi Kırdar City Hospital will create 48 preterm newborns with 28-33 gestation weeks, which are hospitalized between March 2023 and March 2024, which meet the inclusion criteria and received written consent from their parents. Intake swallowing coordination but 32-34. Since it develops after the gestation week, (Törüner ve Büyükgönenç, 2012) sampling will be included in preterm newborns smaller than the 34th gestation week.

Power analysis was performed using the G*Power (v3.1.9.2) program to determine the number of samples. The strength of the study is 1-β (β = II. The probability of type error is expressed as ) and in general research should have 80% power. S. S. Based on the study of Ceylan et al, the effect size of the calculation result made based on the difference of Gastric residuals (ml) measurements according to the supine and right lateral position was calculated as d=0.420 and at the level of α=0.05 %It has been calculated that there must be at least 47 preterm newborns in total to get 80 powers. Considering the loss of case, the number of samples was determined as 48.

Inclusion criteria; The participants who are in the 28-33 gestation week according to the mother's last men's history, are the 1st enteral feeding after mechanical ventilation, fed with breast milk, clinically stable and enteral nutrition, Newborns provided with at least 50% ' of enteral nutrition, fed with free flow and orogastric probe, and received informed consent from parents will be included in the study.

Exclusion criteria; With cerebrovascular disease, with a need for mechanical ventilation, diagnosed with NEC, vomiting, abdominal distension, nasal mechanical obstruction, congenital anomaly, gastrochysis or congenital diaphragm hernia, Newborns with apnea episodes, severe neurological disease will not be included in the study. The participants that worsen clinically after being included in the sample group will be removed from the study.

Independent variables: Positioning (Prone, right lateral and semi-elevated supine position) Dependent variables: Preterm newborn abdominal NIRS value, fractional oxygen extraction value, gastric residual volume.

Research Hypotheses H0: There is no difference between the effects of the three positions on gastric residual volume, abdominal oxygenation, and fractional oxygen extraction.

H1: Abdominal oxygenation and oxygen level (SPO2) are higher in the prone position than in the semi-elevated supine position and the right lateral position.

H2: Abdominal oxygenation and oxygen level (SPO2) are higher in the right lateral position than in the semi-elevated supine position.

H3: The amount of gastric residual volume in the prone position is lower than in the semi-elevated supine position and the right lateral position.

H4: The amount of gastric residual volume in the right lateral position is lower than in the semi-elevated supine position.

H5: Fractional oxygen extraction in the prone position is lower than in the right lateral and semi-elevated supine position.

Data Collection Method The data were collected from Kartal Dr. It will be collected in the neonatal intensive care unit of Lütfi Kırdar City Hospital. Study data will be collected by two investigators. The investigators responsible for the study, the subjects, and the statistician who will analyze the study will be blinded to the data. In the study, the blinding technique was planned as three blinds.

I ntroductory Information and Data Collection Form The intervention group of each participant included in the sample, week of gestation (according to last menstrual period), date, type of delivery, postnatal age, birth weight, postnatal body weight, gender, receiving intravenous fluid support, mean NIRS value, heart rate, and saturation value, amount and color of gastric residual volume before feeding, presence of a disease requiring medical treatment will be recorded.

To assess abdominal oxygenation (ArSO2), the NIRS sensor probe will be placed over the lower abdomen (under the umbilicus) and monitored. The participants who meet the inclusion criteria will be monitored through the NIRS for three feedings. Average NIRS values will be calculated for periods immediately before, during and after feeding. NIRS values will be recorded by the monitor, after the monitoring, the picture of the records will be taken from the monitor. During the follow-up, the location of the probe and the NIRS value will be followed by the investigators who collect data. The probe position will be changed to be in the lower abdomen before each feeding during the follow-up period. While NIRS values are recorded, pulse oximetry values will also be recorded.

Materials to be Used

1. Gastric residual volume Gastric residual volume will be checked manually using a 5 ml syringe prior to feeding. Gastric residue will be excreted or given back in consultation with the doctor according to its amount and color.
2. Breast Milk: Name and date control of the milk stored in milk storage bags in the refrigerator will be made. The breast milk drawn into the injector in accordance with the hygiene rules will be given to the participants after it reaches the appropriate temperature (must be at body temperature) in hot water. Heating breast milk above 40°C is not recommended as it will destroy immunologically active factors.
3. Positioning: Participants will be placed in the supine position during feeding. Feeding will be done every 2-3 hours. Participants will be positioned in one position for 2 hours after feeding.

   * Semi-elevated supine position
   * prone position
   * Right lateral position

Data Collection Feeding time will take 10-20 minutes. The participants will be included in the sampling from their 1st feeding after weaning off the mechanical ventilator. The procedure will begin when participants in all groups are calm. The entire application process will be carried out in the neonatal intensive care unit and all materials will be prepared before the procedure. In all three intervention groups, gastric residue will be checked with a 5 ml injector just before feeding, and the residual content will be discarded or returned with the decision of the doctor. The NIRS sensor probe will be attached to the lower abdomen. Since the cost of the probes is high, reversebl probes will be used and their cleaning will be provided with high-level disinfectant (Ecolab wipes). One NIRS probe will be used for two participants. The same enteral feeding protocol will be applied to all participants. In the institution where the study will be conducted, minimal enteral nutrition is started in participants, with breast milk being the first choice after 24 hours postnatally. Then, if the participant can tolerate enteral feeding, the amount is gradually increased each day. Decisions to increase feeding volume, stop feeding and use breast milk fortifier are made by the clinical team based on local protocols. The amount and frequency of feeding will be decided according to the gestational week, body weight and clinical condition of the participant.

Data Analysis NCSS (Number Cruncher Statistical System) 2020 Statistical Software (NCSS LLC, Kaysville, Utah, USA) program will be used for statistical analysis. While evaluating the study data, Shapiro Wilks test and Box Plot charts will be used to evaluate the conformity of the data to the normal distribution, as well as descriptive statistical methods (mean, standard deviation, median, frequency and ratio). Student's t test in the evaluation of two groups of normally distributed variables; Oneway Anova test will be used in the comparison of three groups and above, and the Bonferroni test will be used to determine the group that causes the difference. Repeated Measures test for evaluations according to three positions within the group; Bonferroni test will be used in post hoc evaluations and Paired Sample t test will be used in peer-to-peer evaluations. Mann Whitney U test in the evaluation of non-normally distributed variables according to two groups; Kruskal Wallis test will be used in the comparison of three groups and above, and Dunn test will be used to determine the group causing the difference. Friedman test post hoc Dunn test in the evaluations according to three positions within the group; Wilcoxon Signed Rank test will be used for peer-to-peer evaluations. Pearson or Spearman's correlation analysis will be used according to the distribution in the evaluation of the relations between the variables; Linear regression models will be made in further evaluations. Chi-square test and Fisher's Exact test will be used in the comparison of qualitative data. The results will be evaluated at the 95% confidence interval, at the p<0.05 level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns who are at 28-33 weeks of gestation according to the last menstrual period of the mother,
* Preterm newborns who are breastfed,
* Preterm newborns who are clinically stable and enteral feeding started,
* Preterm newborns who are first enteral nutrition 24 hours after mechanical ventilation,
* Preterm newborns who are at least 50% of their nutrition provided with enteral nutrition,
* Free Newborns fed by flow and orogastric tube and with informed consent of the parents will be included in the study.

Exclusion Criteria:

* Preterm newborns requiring mechanical ventilation,
* Preterm newborns diagnosed with NEC,
* Preterm newborns vomiting,
* Preterm newborns who have abdominal distension,
* Preterm newborns who have nasal mechanical obstruction,
* Preterm newborns who have congenital anomalies,
* Preterm newborns who have gastrointestinal problems such as gastroschisis or congenital diaphragmatic hernia,
* Preterm newborn who have cerebrovascular disease, apnea episodes, severe neurological disease, were included in the study. will not be included,
* Preterm newborns who worsen clinically after inclusion in the sample group will be excluded from the study.

Ages: 28 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Preterm newborn abdominal NIRS value | Preterm newborns whose feedings are every two hours will be monitored for 6 hours and those whose feedings are every three hours will be monitored for 9 hours. Preterm newborns will be monitored for a total of three feedings
  Average NIRS values will be calculated for periods immediately before, during and after feeding. NIRS values will be recorded by the device, after the monitoring, the picture of the records will be taken from the device.
Fractional oxygen extraction value | Preterm newborns whose feedings are every two hours will be monitored for 6 hours and those whose feedings are every three hours will be monitored for 9 hours. Preterm newborns will be monitored for a total of three feedings
  Pulse oximeter and NIRS monitor will be used together to determine fractional oxygen extraction.
Gastric residual volume | Preterm newborns whose feedings are every two hours will be monitored for 6 hours and those whose feedings are every three hours will be monitored for 9 hours. Preterm newborns will be monitored for a total of three feedings
  Gastric residual volume will be checked manually using a 5 ml syringe prior to feeding. Gastric residue will be excreted or given back in consultation with the doctor according to its amount and color.

CONTACTS AND LOCATIONS:
Locations (1):
- Hande Özgörü, Merkez, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boquien CY. Human Milk: An Ideal Food for Nutrition of Preterm Newborn. Front Pediatr. 2018 Oct 16;6:295. doi: 10.3389/fped.2018.00295. eCollection 2018. PMID 30386758
- [Background] Braski K, Weaver-Lewis K, Loertscher M, Ding Q, Sheng X, Baserga M. Splanchnic-Cerebral Oxygenation Ratio Decreases during Enteral Feedings in Anemic Preterm Infants: Observations under Near-Infrared Spectroscopy. Neonatology. 2018;113(1):75-80. doi: 10.1159/000481396. Epub 2017 Nov 8. PMID 29131125
- [Background] Barsan Kaya T, Aydemir O, Tekin AN. Prone versus supine position for regional cerebral tissue oxygenation in preterm neonates receiving noninvasive ventilation. J Matern Fetal Neonatal Med. 2021 Oct;34(19):3127-3132. doi: 10.1080/14767058.2019.1678133. Epub 2019 Oct 15. PMID 31615310
- [Background] Chen SS, Tzeng YL, Gau BS, Kuo PC, Chen JY. Effects of prone and supine positioning on gastric residuals in preterm infants: a time series with cross-over study. Int J Nurs Stud. 2013 Nov;50(11):1459-67. doi: 10.1016/j.ijnurstu.2013.02.009. Epub 2013 Mar 26. PMID 23537895
- [Background] Corvaglia L, Martini S, Battistini B, Rucci P, Aceti A, Faldella G. Bolus vs. continuous feeding: effects on splanchnic and cerebral tissue oxygenation in healthy preterm infants. Pediatr Res. 2014 Jul;76(1):81-5. doi: 10.1038/pr.2014.52. Epub 2014 Apr 8. PMID 24713819
- [Background] Corvaglia L, Martini S, Battistini B, Rucci P, Faldella G, Aceti A. Splanchnic Oxygenation at First Enteral Feeding in Preterm Infants: Correlation With Feeding Intolerance. J Pediatr Gastroenterol Nutr. 2017 Apr;64(4):550-554. doi: 10.1097/MPG.0000000000001308. PMID 27467111
- [Background] Cortez J, Makker K, Kraemer DF, Neu J, Sharma R, Hudak ML. Maternal milk feedings reduce sepsis, necrotizing enterocolitis and improve outcomes of premature infants. J Perinatol. 2018 Jan;38(1):71-74. doi: 10.1038/jp.2017.149. Epub 2017 Sep 28. PMID 29048409
- [Background] Ceylan SS, Keskin Z. Effects of two different positions on stress, pain and feeding tolerance of preterm infants during tube feeding. Int J Nurs Pract. 2021 Oct;27(5):e12911. doi: 10.1111/ijn.12911. Epub 2020 Dec 9. PMID 33300212
- [Background] da Costa CS, Greisen G, Austin T. Is near-infrared spectroscopy clinically useful in the preterm infant? Arch Dis Child Fetal Neonatal Ed. 2015 Nov;100(6):F558-61. doi: 10.1136/archdischild-2014-307919. Epub 2015 Jul 27. PMID 26215405
- [Background] Demirel G, Oguz SS, Celik IH, Erdeve O, Dilmen U. Cerebral and mesenteric tissue oxygenation by positional changes in very low birth weight premature infants. Early Hum Dev. 2012 Jun;88(6):409-11. doi: 10.1016/j.earlhumdev.2011.10.005. Epub 2011 Nov 15. PMID 22088784
- [Background] Dani C, Coviello C, Montano S, Remaschi G, Petrolini C, Strozzi MC, Maggiora E, Sabatini M, Gazzolo D. Effect on splanchnic oxygenation of breast milk, fortified breast milk, and formula milk in preterm infants. Pediatr Res. 2021 Jan;89(1):171-174. doi: 10.1038/s41390-020-0935-1. Epub 2020 May 7. PMID 32380507
- [Background] Garvey AA, Dempsey EM. Applications of near infrared spectroscopy in the neonate. Curr Opin Pediatr. 2018 Apr;30(2):209-215. doi: 10.1097/MOP.0000000000000599. PMID 29369068
- [Background] Goldshtrom N, Isler JR, Sahni R. Comparing liver and lower abdomen near-infrared spectroscopy in preterm infants. Early Hum Dev. 2020 Dec;151:105194. doi: 10.1016/j.earlhumdev.2020.105194. Epub 2020 Sep 17. PMID 33017708
- [Background] Hay WW Jr, Hendrickson KC. Preterm formula use in the preterm very low birth weight infant. Semin Fetal Neonatal Med. 2017 Feb;22(1):15-22. doi: 10.1016/j.siny.2016.08.005. Epub 2016 Aug 30. PMID 27595621
- [Background] Liao SM, Rao R, Mathur AM. Head Position Change Is Not Associated with Acute Changes in Bilateral Cerebral Oxygenation in Stable Preterm Infants during the First 3 Days of Life. Am J Perinatol. 2015 Jun;32(7):645-52. doi: 10.1055/s-0034-1390348. Epub 2014 Oct 5. PMID 25282608
- [Background] Martini S, Aceti A, Beghetti I, Faldella G, Corvaglia L. Feed-related Splanchnic Oxygenation in Preterm Infants With Abnormal Antenatal Doppler Developing Gut Complications. J Pediatr Gastroenterol Nutr. 2018 May;66(5):755-759. doi: 10.1097/MPG.0000000000001804. PMID 29112084
- [Background] Ozdel D, Sari HY. Effects of the prone position and kangaroo care on gastric residual volume, vital signs and comfort in preterm infants. Jpn J Nurs Sci. 2020 Jan;17(1):e12287. doi: 10.1111/jjns.12287. Epub 2019 Oct 23. PMID 31642602
- [Background] Patel AK, Lazar DA, Burrin DG, Smith EO, Magliaro TJ, Stark AR, Brandt ML, Zamora IJ, Sheikh F, Akinkuotu AC, Olutoye OO. Abdominal near-infrared spectroscopy measurements are lower in preterm infants at risk for necrotizing enterocolitis. Pediatr Crit Care Med. 2014 Oct;15(8):735-41. doi: 10.1097/PCC.0000000000000211. PMID 25068253
- [Background] Parker L, Torrazza RM, Li Y, Talaga E, Shuster J, Neu J. Aspiration and evaluation of gastric residuals in the neonatal intensive care unit: state of the science. J Perinat Neonatal Nurs. 2015 Jan-Mar;29(1):51-9; quiz E2. doi: 10.1097/JPN.0000000000000080. PMID 25633400
- [Background] Singh B, Rochow N, Chessell L, Wilson J, Cunningham K, Fusch C, Dutta S, Thomas S. Gastric Residual Volume in Feeding Advancement in Preterm Infants (GRIP Study): A Randomized Trial. J Pediatr. 2018 Sep;200:79-83.e1. doi: 10.1016/j.jpeds.2018.04.072. Epub 2018 Jun 1. PMID 29866595
- [Background] Seager E, Longley C, Aladangady N, Banerjee J. Measurement of gut oxygenation in the neonatal population using near-infrared spectroscopy: a clinical tool? Arch Dis Child Fetal Neonatal Ed. 2020 Jan;105(1):76-86. doi: 10.1136/archdischild-2018-316750. Epub 2019 Jun 1. PMID 31154420
- [Background] Tran NN, Kumar SR, Hodge FS, Macey PM. Cerebral Autoregulation in Neonates With and Without Congenital Heart Disease. Am J Crit Care. 2018 Sep;27(5):410-416. doi: 10.4037/ajcc2018672. PMID 30173174
- [Background] Ziehenberger E, Urlesberger B, Binder-Heschl C, Schwaberger B, Baik-Schneditz N, Pichler G. Near-infrared spectroscopy monitoring during immediate transition after birth: time to obtain cerebral tissue oxygenation. J Clin Monit Comput. 2018 Jun;32(3):465-469. doi: 10.1007/s10877-017-0052-9. Epub 2017 Aug 19. PMID 28823017